CLINICAL TRIAL: NCT02876991
Title: Evaluation of Sodium Fluoride PET in the Identification of Bone Metastases in Patients Having Undergone a Choline PET for Occult Recurrence of Prostatic Adenocarcinoma
Acronym: FNa-CHOLINE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015-A00021-48
Record Dates: First submitted 2016-08-10; First posted 2016-08-24 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Bone Metastasis
Keywords: choline positron emission tomography; occult recurrence; prostatic adenocarcinoma; sodium fluoride positron emission tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sodium fluoride PET (Other): Before inclusion, patients undergo choline PET to assess an occult recurrence of prostate cancer.
  After inclusion, they undergo sodium fluoride PET.
  Interventions: Procedure: Sodium fluoride PET

INTERVENTIONS:
Procedure: Sodium fluoride PET — Sodium fluoride Pet is realized maximum after 4 weeks from choline PET (inclusion).
  Injection of 4MBq 18F-FNa/kg of body weight is followed after 60 min (± 5 min) by acquisition of images on Biograph 6 PET/CT scanner (SIEMENS).
  Data from sodium fluoride PET are interpreted independently and blind from other data by 3 medical doctors (2 at hospital of Nancy and 1 at hospital of Strasbourg) (for inter-judge reproducibility); a second interpretation of data is consensually realized by 2 of 3 readers, limited to discordant analyses (metastatic status or not, and/or number of lesions); results from this second interpretation are final results.

SUMMARY:
The purpose is to evaluate if sodium fluoride PET in patients having already undergone a choline PET negative for bone extension (non-metastatic status) modifies the status of patients concerning the existence or not of bone metastases.

Secondary purposes are:

* To evaluate if detection of bone metastasis by sodium fluoride PET, not detected by choline PET, leads to change of treatment
* To evaluate inter-technique concordance (choline vs sodium fluoride PET) of results (metastatic status and number of lesions)
* To evaluate the inter-judge concordance of interpretation of sodium fluoride PET
* To study the discordance of metastatic status of 2 techniques.

ELIGIBILITY:
Inclusion Criteria:

* Prostate adenocarcinoma regardless of Gleason score
* Patients having undergone radical treatment (prostatectomy or radiotherapy (external or brachytherapy) +/- conco-adjuvant hormonal therapy)
* Level of Prostate Specific Antigen (PSA) indicating recurrence: PSA > 0.2 ng/ml in case of prostatectomy (in 2 consecutive tests in less than 1 month) or elevation of PSA of at least 2 ng/ml above nadir in case of radiotherapy or brachytherapy (in 2 consecutive tests in less than 1 month)
* Negative conventional assessment (thoracic-abdominal-pelvic scanner and bone scintigraphy) during 6 weeks before inclusion
* Patient having undergone a choline PET at CHRU Nancy
* Signed informed consent
* Affiliation to French social security
* Absence of contraindications to sodium fluoride PET

Exclusion Criteria:

* Refusal or impossibility of informed consent
* Patient incapable to consent
* Patient deprived of liberty
* Person under legal protection
* Person in life-and-death emergency
* Drug addiction, alcoholism, psychological problems affecting patient compliance
* Severe co-morbidities
* Modification of hormonal therapy (if applicable) during 3 months before inclusion
* Renal insufficiency (creatinine clearance < 60 ml/min) detected during last assessment before inclusion
* Other progressive tumors (recovered cancers are not a non-inclusion criteria)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2016-02; Primary Completion 2018-08 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with choline PET negative and sodium fluoride PET positive for bone extension (metastasis) | Execution of sodium fluoride PET (up to 4 weeks from choline PET; from baseline up to 4 weeks)

SECONDARY OUTCOMES:
Inter-strategy concordance of diagnosis evaluated by kappa coefficient | Execution of sodium fluoride PET (up to 4 weeks from choline PET; from baseline up to 4 weeks)
  Concordance between results of choline PET and sodium fluoride PET
Metastatic status and number of lesions detected respectively by sodium fluoride PET and choline PET | Execution of sodium fluoride PET (up to 4 weeks from choline PET; from baseline up to 4 weeks)
Metastatic status and number of lesions identified by 3 medical doctors of 2 different centres in sodium fluoride PET | Execution of sodium fluoride PET (from baseline up to 4 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre OLIVIER, Pr, Principal Investigator — Service de Médecine Nucléaire - CHRU de Nancy-Brabois - Vandœuvre-lès-Nancy
Locations (1):
- Service de Médecine Nucléaire CHRU de Nancy-Brabois, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No